CLINICAL TRIAL: NCT04473547
Title: Adherence of Nursing Students to Preventive Measures Towards Coronavirus Disease 19 During Written Exams
Brief Title: COVID 19 Preventive Measures Among Mansoura Nursing Students
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, mohamed elsayed hamed elzeky, lecturer-medical surgical nursing department-faculty of nursing mansoura university, Mansoura University
Other Study IDs: p.0203
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: COVID 19; preventive measures; nursing students
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to identify nursing students knowledge gaps, risk perceptions and adherence to COVID 19 preventive measures during written exam period and In addition due to the possibility of being infected with COVID-19 during exams this study will evaluate covid-19 symptoms rate during exam period and factors affecting its development .

DETAILED DESCRIPTION:
As of june,27,2020, Egypt lift most COVID-19 restrictions and government decided to held written exams for final year students with precautionary measures. Students reported fears regarding the possibility of being infected during exams period and want to postpone or cancel exams due to possible contact during transportation and meeting in classes. Education have been provided to population in general and students in special through social media, social networks, community leaders to take precautionary measures during exams.

Studies provide support for the notion of increased vulnerability to respiratory tract infections with exposure to psychological stress . one of specific stress is Academic Exam stress that has been linked with immuno-suppression.

Exams are stressful experience and a place for student gathering , moreover there is no research about adherence level or factors affecting adherence to COVID-19 precautions among nursing students during exam period. Nursing students are future professionals who can address new emerging infectious diseases.

the study aims to analyze students adherence to COVID 19 preventive measures and to to identify the knowledge gaps, risk perceptions and factors affecting students adherence which could guide the design of better nursing education curricula regarding COVID-19 as a preparation for final year nursing students to internship year which will be on September 2020 . In addition due to the possibility of being infected with COVID-19 during exams or during their internship year this study will evaluate covid-19 symptoms rate during exam period and factors affecting its development .

ELIGIBILITY:
Inclusion Criteria:

* Students who agree to participate.
* Students of both gender .
* Students who have access to internet and have whatsapp account

Exclusion Criteria:

* Students diagnosed with COVID-19 before.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A convenient sample of 215 4th level 2nd term bachelor nursing students undergoing written exam in July period and agree to participate in study will be involved. The target population are 484 students who are undergoing written exam this year. The required sample size was calculated by Raosoft sample size calculator. Based on the estimated population and response distribution of 50%, the required sample size is 215 with a confidence level of 95% and 5% margin of error.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
adherence level to coronavirus disease 19 preventive measures among nursing students during written exams. | from 15\7\2020 to 1\8\2020
  an online questionnaire consists of six sections as following (hand hygiene practices, social distancing, respiratory hygiene, social distancing, cleaning and disinfection and nurse role model. Each item will be answered as "always" or "sometimes" or " rarely" or "never" .
number of students who develop possible covid-19 symptoms during written exams | longitudinal over 6 weeks from 15\7\2020 to 30\8\2020
  Online questionnaire will be sent to students every 2 weeks for 6 weeks (during and after exam period by two weeks )asking about the appearance of new symptoms of COVID-19 including ( fever, dry cough, shortness of breath, new loss of taste or smell, muscle pain, …) every two weeks.
Eye,nose,mouth,Face and mask touch frequency during written exams | from 15\7\2020 to 1\8\2020
  students will be videotaped during exams and analyzed using observational checklist for hand to eye , nose, mouth, mask and face touch frequency

SECONDARY OUTCOMES:
nursing students knowledge level of COVID 19 | from 15\7\2020 to 30\8\2020
  A correct answer will be scored (1) while incorrect or missed answer will be scored (0). The level of knowledge will be considered poor if the percentage mean score is less than 50%, fair if from 50 to less than 75%, and good if more than or equal 75% .
COVID 19 risk perception level among nursing students undergoing written exams | from 15\7\2020 to 30\8\2020
  Each item will be answered as "no" (0) or "not sure" (1) or" yes" (2). A high score meant a high risk perception.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided